CLINICAL TRIAL: NCT00751933
Title: A Controlled Study of Salmonella Ty21a and Cholera/ ETEC-vaccine and the Role of Oats in Daily Diet as a New Treatment in Patients With Mild or Moderate Ulcerative Colitis.
Brief Title: Vaccines and Dietary Oats in the Treatment of Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of patients compatible with the protocol´s criteria
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Vest (Other)
Responsible Party: Principal Investigator, Gunnar Nysæter, Senior Consultant, Haukeland University Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 16816 NSD; 2007-002415-88 (SLV/EudraCT) (Other: Statens Legemiddelverk); 911305 (Helse Vest RHF) (Other: Helse Vest RHF); 82/2007 (P REK Nord) (Other: Regional Etisk Komite); 16816 (NSD) (Other: Norsk Samfunnsvitenskapelig Datatjeneste)
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Results first posted 2015-04-28 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; Vaccines; Oats
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Ty21a typhoid vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2 (Experimental): Vaccination with Vivotif and Dukoral
  Interventions: Biological: Vaccine Vivotif + Vaccine Dukoral
- 3 (Experimental): Dietary supplement with oats
  Interventions: Dietary Supplement: Oats
- 4 (Placebo Comparator): Placebo instead of vaccines No dietary supplement
  Interventions: Other: Placebo
- 1 (Experimental): Vaccination with Vivotif and Dukoral + dietary supplement with oats.
  Interventions: Biological: Vaccine Vivotif + Vaccine Dukoral + oats

INTERVENTIONS:
Biological: Vaccine Vivotif + Vaccine Dukoral + oats — Vivotif 1 capsule at study day 1,3,5 and 7. Dukoral oral mixture taken with sodium hydrogen carbonate in water at study day 1 and 14.
  One daily portion of oats porridge made from oats grain 1dL and water, 6 days a week for 6 months.
  Other Names: Ty21a; Vibrio cholera O1 Ogawa, inactivated
  Arms: 1
Biological: Vaccine Vivotif + Vaccine Dukoral — Vivotif 1 capsule at study day 1,3,5 and 7. Dukoral oral mixture taken with sodium hydrogen carbonate in water at study day 1 and 14.
  Other Names: Ty21a; Vibrio cholera O1 Ogawa, inactivated
  Arms: 2
Dietary Supplement: Oats — One daily portion of oats porridge made from oats grain 1dL and water, 6 days a week for 6 months.
  Arms: 3
Other: Placebo — Placebo capsules instead of Vivotif capsules Placebo mixture instead of liquid Dukoral vaccine
  Arms: 4

SUMMARY:
Ulcerative colitis is a chronic inflammatory bowel disease caused by an imbalance between natural defence mechanisms in the intestinal mucosa and microbes in the intestinal lumen. We hypothesise that an improvement or even normalisation of this balance may be achieved by the use of vaccines and dietary oats. The combined use of oral typhoid vaccine and cholera/ETEC-vaccine is supposed to stimulate mucosal defence factors, while dietary oats modifies the microbial environment inside the intestinal lumen. Or study aim is to show if such treatment brings symptom relief to patients with ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* ulcerative colitis of at least 4 months duration
* disease activity index score (Walmsley) >5 and </=13
* patients taking no ulcerative colitis relevant medicine, or stable doses of aminosalicylates or maximum 10mg prednisolon daily the last 2 weeks before study entry. They must remain on the same dose throughout the study (6 months).
* stool examination negative for enteric pathogens, clostridium difficile toxin and parasites

Exclusion Criteria:

* ulcerative colitis disease activity index >13
* symptoms of bowel obstruction
* other serious medical condition
* use of any of the study vaccines during the last two years
* use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first vaccine dose, or planned use during study period
* pregnant or planning to become pregnant
* breastfeeding
* chronic administration of prednisolone more than 10mg per day or steroids of equivalent dose the last 2 weeks before the first vaccine dose
* treatment with anti-tumor necrosis factor within 3 months prior to the first vaccine dose
* use of other immunosuppressants or immune modifying drugs within 30 days prior to the first vaccine dose

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Nysæter, MD, Principal Investigator — Department of Medicine,Haukeland University Hospital, Bergen, Norway
Locations (1):
- Department of Medicine, Haukeland Universtiy Hospital, Bergen, Norway

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaccine Arm 2: Vaccination with Vivotif and Dukoral
  Vaccine Vivotif + Vaccine Dukoral: Vivotif 1 capsule at study day 1,3,5 and 7. Dukoral oral mixture taken with sodium hydrogen carbonate in water at study day 1 and 14.
- Oats Supplement 3: Dietary supplement with oats
  Oats: One daily portion of oats porridge made from oats grain 1dL and water, 6 days a week for 6 months.
- Placebo 4: Placebo instead of vaccines No dietary supplement
  Placebo: Placebo capsules instead of Vivotif capsules Placebo mixture instead of liquid Dukoral vaccine
- Vaccine and Oats 1: Vaccination with Vivotif and Dukoral + dietary supplement with oats.
  Vaccine Vivotif + Vaccine Dukoral + oats: Vivotif 1 capsule at study day 1,3,5 and 7.
  Dukoral oral mixture taken with sodium hydrogen carbonate in water at study day 1 and 14.
  One daily portion of oats porridge made from oats grain 1dL and water, 6 days a week for 6 months.
Period: Overall Study
Arm/Group | Vaccine Arm 2 | Oats Supplement 3 | Placebo 4 | Vaccine and Oats 1
Started | 0 | 1 | 1 | 1
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Arms: Three patients entered the study, one man, two women. Age 24-41 years. The study was terminated due to lack of patients for inclusion.
Arm/Group | All Arms
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 32 [24 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Region of Enrollment [Number; unit: participants]
  Norway | 3

OUTCOME MEASURES:

1. Primary Outcome: Symptom Score Improvement of 3 or More During or After 6 Months
Description: No patient completed the study, therefore we have no information to report.
Time Frame: 6 months
Groups:
- All Arms: No patient completed the study, therefore we have no information to report.
Arm/Group | All Arms
Number analyzed (Participants) | 0

2. Secondary Outcome: Symptom Score Improvement of 2 or More During or After 6 Months
Description: No patient completed the study, therefore we have no information to report.
Time Frame: 6 months
Arm/Group | All Arms
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- All Arms: No adverse effects were recorded.
Arm/Group | All Arms
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes